CLINICAL TRIAL: NCT00002635
Title: PHASE II TRIAL OF 9-AMINOCAMPTOTHECIN IN ADVANCED CUTANEOUS T CELL LYMPHOMA
Brief Title: Aminocamptothecin in Treating Patients With T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000064085; YALE-HIC-7862; NCI-T94-0189D
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2001-03

CONDITIONS: Lymphoma
Keywords: stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: filgrastim
Drug: aminocamptothecin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of aminocamptothecin in treating patients with advanced cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity of aminocamptothecin (9-AC) administered by 72-hour infusion in patients with advanced cutaneous T-cell lymphoma. II. Assess the toxic effects of 9-AC administered on this schedule.

OUTLINE: Single-Agent Chemotherapy. Aminocamptothecin, 9-AC, NSC-603071.

PROJECTED ACCRUAL: A total of 30 patients will be accrued; if no more than 1 response is seen in the first 15 patients, the study will close. Probable duration of study is 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, advanced stages IIB/III/IV cutaneous T-cell lymphoma Measurable or evaluable disease required Measurable disease includes: Skin disease evaluated by clinical assessment grid method Lesion measurable on imaging (i.e., CT measurement of lymph nodes) Pure osteolytic lesion Unidimensional lesion for which a normal measurement is available (e.g., mediastinal width on x-ray) Evaluable disease defined as malignant disease evident on physical or radiographic exam but not measurable by ruler or caliper, i.e.: Pelvic masses Confluent multinodular lung metastases Skin metastases CNS metastases eligible if stable for at least 4 weeks following completion of surgery or radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: ANC at least 1,500 Platelets at least 100,000 Hepatic: Bilirubin no greater than 1.5 mg/dL AST less than 3 times normal Renal: Creatinine no greater than 1.5 mg/dL Other: No contraindication to indwelling central venous catheter No active infection including HIV No other medical condition that would preclude protocol compliance No pregnant or nursing women Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior biological therapy allowed Chemotherapy: Prior systemic chemotherapy allowed Patients with more than 1 prior regimen analyzed separately At least 4 weeks since chemotherapy (6 weeks since nitrosoureas or mitomycin) Endocrine therapy: Not specified Radiotherapy: Prior skin irradiation allowed At least 4 weeks since wide-field radiotherapy Surgery: Fully recovered from prior surgery Other: Prior topical therapy allowed Prior PUVA allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1995-05; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Murren, MD, Study Chair — Yale University
Locations (3):
- United States (3):
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - New England Medical Center Hospital, Boston, Massachusetts